CLINICAL TRIAL: NCT06324773
Title: Prevalence of Postpartum Family Planning Uptake and Its Association With Joint Spousal Decision-Making in Family Planning: A Community-Based Cross-Sectional Study in Rural Sindh, Pakistan
Brief Title: Prevalence of Postpartum Family Planning and Its Association With Spousal Joint Decision-Making in Family Planning
Status: Completed | Type: Observational
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Shiyam Sunder, MBBS, MSc, Principal Investigator, Aga Khan University
Other Study IDs: 9867
Record Dates: First submitted 2024-03-12; First posted 2024-03-22 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Postpartum Family Planning

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This community-based cross-sectional study investigates the prevalence of postpartum family planning (PPFP) uptake and its association with joint spousal family planning decision-making among married women in rural Sindh, Pakistan. The study, conducted in Thatta District with a population of approximately 0.98 million people, addresses sociodemographic challenges including high fertility rates, maternal and newborn mortality, and low contemporary contraception use. Targeting married women aged 18-49 who gave birth within the past year, the research utilizes data from the Global Network's Maternal and Newborn Health Registry. Data collection involves a pretested questionnaire administered by trained female data collectors. Statistical analysis includes descriptive statistics and logistic regression using STATA 17. The study aims to fill knowledge gaps regarding factors influencing PPFP uptake, particularly the role of joint decision-making in family planning. Findings could inform targeted interventions to enhance maternal and child health, contribute to existing knowledge, and guide policymakers and healthcare providers in addressing the unmet need for family planning in rural Pakistan.

ELIGIBILITY:
Inclusion Criteria:

* Women who are married and gave birth a year ago
* Living within the Maternal Neonatal Health Registry catchment area for at least one year.
* Women who will give their consent.

Exclusion Criteria:

* Pregnant women.
* Women who are critically ill and who face significant cognitive barriers that hinder their understanding and participation in the study.

Ages: 15 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Married women of reproductive age (18-49) who gave birth a year ago and registered in the Maternal and Newborn Health Registry in Thatta District Sindh, Pakistan.
Sampling Method: Probability Sample
Enrollment: 524 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of Postpartum Family Planning Uptake | In past one year
  Number of women who utilized postpartum family planning.
Frequency of spousal joint decision making for uptake of postpartum family planning | In past one year
  The outcome measures the frequency at which spouses make joint decisions regarding the uptake of postpartum family planning methods
Comparison between spousal joint decision making is using postpartum family planning method and non-users. | in past one year
  Compare spousal joint decision-making in couples using postpartum family planning methods versus those not using them.

CONTACTS AND LOCATIONS:
Locations (1):
- Thatta, Thatta, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khurram J, Hasnani FB, Saleem S, Tikmani SS. Prevalence of postpartum family planning uptake and its association with couples' joint decision-making: a community-based cross-sectional study in rural Sindh, Pakistan. BMJ Public Health. 2025 Dec 21;3(2):e002982. doi: 10.1136/bmjph-2025-002982. eCollection 2025. PMID 41431612